CLINICAL TRIAL: NCT04972071
Title: Multi-Centre Cluster-Randomized Implementation of Canadian Syncope Risk Score Based Practice Recommendations for Emergency Department Syncope Management
Brief Title: SW-RCT Implementation of Canadian Syncope Risk Score Based Practice Recommendations
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ottawa Hospital Research Institute (Other)
Responsible Party: Principal Investigator, Venkatesh Thiruganasambandamoorthy, Professor and Senior Scientist, Ottawa Hospital Research Institute
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 3371
Record Dates: First submitted 2021-07-12; First posted 2021-07-22 (Actual); Last update posted 2025-03-27 (Actual); Status verified 2025-03

CONDITIONS: Syncope
Keywords: Syncope; Emergency Department; Risk Stratification
MeSH Terms: conditions — Syncope; Emergencies

STUDY DESIGN:
Intervention Model Description: A Stepped Wedge-Controlled Randomized Trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- CSRS practice recommendation (Other): Knowledge translation of the Canadian Syncope Risk Score (CSRS) based practice recommendations
  Interventions: Other: Knowledge translation (KT) of the CSRS based practice recommendations

INTERVENTIONS:
Other: Knowledge translation (KT) of the CSRS based practice recommendations — The components of the practice recommendations include: 1) evidence-informed systematic clinical evaluation with appropriate history, physical examination and in-ED investigations (e.g., troponin testing, work-up for pulmonary embolism and CT head) for detecting serious underlying conditions and predicting 30-day serious outcomes; 2) application of the CSRS for risk-stratification at the end of ED visit after no serious underlying conditions for the syncope were identified; 3) use of patient information materials to aid in disposition; and 4) the use of 15-day outpatient cardiac monitoring for CSRS medium and high-risk patients upon ED discharge. All the components of the practice recommendations will be applied by the ED physician treating the patient.

SUMMARY:
Syncope is a common reason for emergency department (ED) presentation. While often benign, some patients have serious and life-threatening underlying causes, both cardiac and non-cardiac, which may or may not be apparent at the time of the initial ED assessment. Identifying which patients will benefit from further investigation, ongoing monitoring and/or hospital admission is essential to reduce both adverse outcomes and high costs. The research team has spent over a decade developing the evidence base for a risk stratification tool directed at optimizing the accuracy of ED decisions: the Canadian Syncope Risk Score (CSRS). This tool is now ready for the final phase of its introduction into clinical practice, namely a robust, multicentre implementation trial of the CSRS-based practice recommendations to demonstrate its real-world effectiveness. These recommendations, if applied, could lead to reduction in hospitalization with only 6% of high-risk patients requiring hospitalization, shorter ED lengths of stay for the 76% of ED syncope patients who are at low risk for 30-day serious outcomes, and more standardized disposition decisions, specifically discharge of 18% of medium-risk patients after appropriate discussion. Hence, the investigators hypothesize that an important reduction in hospitalization and ED disposition time can be achieved by implementing the CSRS-based recommendations with potential improvements in patient safety. The overall objective of this study is to evaluate the effectiveness of the knowledge translation (KT) of the CSRS-based practice recommendations in multiple Canadian EDs using a stepped wedge cluster randomized trial (SW-CRT) on health care efficiency and patient safety.

DETAILED DESCRIPTION:
The investigators will conduct a SW-CRT involving 16 participating ED clusters across Canada. The design will be a batched SW-CRT with two batches of 8 cluster EDs with the first 8 cluster EDs that are ready for the trial included in the first batch. Some EDs will be grouped to avoid contamination between multiple sites operating within the same hospital organization. The total study duration is 16 months for each batch. All clusters in the two batches will start the trial in a control period (usual care) for three months with no intervention being delivered at any site, then sequentially cross over from the control period to the intervention period in random sequence, with 2 clusters crossing over every third month, until all sites have adopted the intervention. Clusters will be randomly allocated to one of four steps (two clusters per step) with step lengths of three months. The first month after crossing over will be designated as a transition period to allow the intervention to be fully implemented. During the first three months of the study, all clusters will be in the control period and during the last three months all clusters will be in the intervention period. Hence, the total study period will be 16 months for each batch.

The following principal research questions will be addressed 1) What is the effect of the knowledge translation and implementation of the CSRS-based practice recommendations on health resource utilization? The health resource utilization measures include the proportion hospitalized, the proportion investigated in the ED, and ED disposition time 2) How and why did the implementation achieve the observed effect? The embedded process evaluation measures align with the RE-AIM (Reach Effectiveness Adoption Implementation Maintenance) framework and include: a) adoption - the proportion of physicians who attended the educational sessions and the proportion who adopted the CSRS in practice; b) reach- the proportion of eligible patients for whom the CSRS was utilized during their ED visit; c) intervention fidelity - the proportion of patients for whom the resulting CSRS recommendations were followed d) maintenance- whether observed adoption rates remain stable or increase over time. 3) What is the effect of the knowledge translation strategy on patient safety, as measured by 30-day serious outcome identification, 30-day and 1-year return ED visits, hospitalizations, and mortality? and 4) validate the ultra-low-risk criteria in a new cohort of patients and assess if the CSRS can be improved in its ability to predict 30-day serious outcomes.

ELIGIBILITY:
Physicians:

Inclusion criteria:

* ED physicians involved in ED syncope care
* Non-ED physicians involved in ED syncope care
* Physician's delegates involved in ED syncope care

Exclusion criteria:

* ED physicians not involved in ED syncope care
* Non-ED physicians not involved in ED syncope care
* Physician's delegates not involved in ED syncope care

Patients:

Inclusion criteria:

* Patients who are adults (aged > 18 years)
* Patients who present to the ED within 24 hours of syncope.

Exclusion criteria:

* Patients who do not fulfill the definition of syncope, namely those with a prolonged loss of consciousness (i.e., > 5 minutes), Glasgow Coma Scale < 15 in patients without dementia (or a change in the mental status from baseline in those with dementia);
* Patients with witnessed obvious seizure, or head trauma preceding the loss of consciousness; and those who are unable to provide proper details (e.g., alcohol intoxication or other substance use).
* Patients who had a serious underlying for the syncope identified during the index ED evaluation and those who were consulted to an inpatient service or hospitalized for reasons other than syncope workup (e.g., social reasons such as inability to cope at home, pain due to the fall, significant trauma).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14400 (Estimated)
Dates: Start 2023-09-18 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Rate of hospitalization | At time of ED disposition, an average timeframe is 6 hours
  to assess the impact on hospital admission

SECONDARY OUTCOMES:
ED disposition time | At time of ED disposition, an average timeframe is 6 hours
  The ED disposition time is defined as the time interval between ED physician initial assessment and ED disposition. We chose this time interval rather than ED length of stay which is the time interval between ED arrival/registration and departure from the ED. The ED disposition time more accurately reflects the active phase of ED physician care for collecting clinical information, work-up of patients and resolution of diagnostic uncertainty. The longer interval of ED length of stay includes wait times both before and after, which are often determined by triage acuity as well as extraneous system factors (e.g., ED and hospital crowding, staffing patterns, sudden influx of patients, availability of inpatient beds and overcapacity protocols, and availability of transportation for a subgroup of patients for whom a decision to discharge has been made);
All-cause mortality | within 30-days and 1-year of the index ED visit
  To assess mortality within 30-days and 1-year of the index ED visit
Number of return ED visits | within 30-days and 1-year
  To assess return ED visits within 30-days and 1-year of the index ED visit
Rate of consultation | 1-year from the index ED visit
  To assess the effectiveness of intervention on consultation performed in the ED
Rate of adoption | Before ED disposition, average of 6 hours
  To assess the adoption of CSRS practice recommendation
Rate of adherence | Before ED disposition, average of 6 hours
  To assess the adherence of the CSRS practice recommendation in the ED
Rate of acceptability | Before ED disposition, average of 6 hours
  To assess the acceptability of the CSRS practice recommendation in the ED

CONTACTS AND LOCATIONS:
Overall Officials: Venkatesh Thiruganasambandamoorthy, CCFP-EM, MSc, Principal Investigator — Ottawa Hospital Research Institute
Locations (15):
- Canada (15):
  - Foothills Medical Centre, Calgary, Alberta
  - St. Boniface Hospital, Winnipeg, Manitoba
  - Health Sicence North, Greater Sudbury, Ontario
  - Hawkesbury and District General Hospital, Hawkesbury, Ontario
  - London Health Sciences Centre, London, Ontario
  - North Bay Regional Health Centre, North Bay, Ontario
  - Thunder Bay Regional Health Sicences Centre, Thunder Bay, Ontario
  - University Health Network, Toronto, Ontario
  - Niagara Health, Welland, Ontario
  - Winchester District Memorial Hospital, Winchester, Ontario
  - Jewish General Hospital, Montreal, Quebec
  - Royal Victoria Hospital & Montreal General Hospital, Montreal, Quebec
  - Centre hospitalier de l'Université Laval, Québec, Quebec
  - Hotel Dieu Hospital of Lévis, Québec, Quebec
  - Hôpital de L'Enfant-Jésus, Québec, Quebec

IPD SHARING:
Plan to Share IPD: No
No plan to share IPD